CLINICAL TRIAL: NCT02789566
Title: Phase 1, Open-Label Study to Evaluate Potential Pharmacokinetic of Orally Administered Primaquine in Healthy Obese Thai Adult Subjects
Brief Title: Pharmacokinetic Study of Primaquine in Healthy Obese Thai Adult Subjects
Acronym: PQ in Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TMEC 11-010
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Obese
Keywords: Primaquine; Pharmacokinetic
MeSH Terms: conditions — Obesity | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regimen (Experimental): Primaquine (PQ) 30 mg base single dose
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Primaquine 30 mg taken after meal in the morning.

SUMMARY:
The primary objective of this study is to provide a description of the pharmacokinetic properties of primaquine and metabolites and characterize these in healthy obese Thai subjects.

This is an open-label, single dose pharmacokinetic study in 10 healthy obese G6PD normal, subjects will be admitted as inpatient to receive 1 regimen for 1 visit only.

DETAILED DESCRIPTION:
Subjects will have 1 hospitalization. The visit will require hospitalization for about 24 hours. After the screening (visit 1), the subject will receive Primaquine (PQ) 30 mg base single dose at first admission (visit 2). Assessment of the safety profile will be done after admission by the investigating team before proceeding to the regimen.

The study will enroll 10 healthy obese subjects (Body mass index [BMI] ≥30 kg/m2) both male and female, age 18-60 years, from the pharmacokinetic unit at Faculty of Tropical Medicine, Mahidol University. Participants will be healthy HIV-1, hepatitis B and C uninfected individuals who comprehend the purpose of the study and have provided written consent. Participants will be screened and eligibility will be based on inclusion and exclusion criteria. If all doses are completed without replacement of subjects, the total number of subjects in this study is 10. All subjects will undergo screening assessments within 7 days prior to the single dose to determine their eligibility for enrollment into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females aged between 18 years to 60 years.
3. BMI ≥ 30 kg/m2 (BMI= body weight[BW](kg)/height(m2))
4. A female is eligible to enter and participate in this study if she is:

   * childbearing potential, has a negative serum pregnancy test at screening and urine pregnancy test prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Read, comprehend, and write at a sufficient level to complete study-related materials.
7. Provide a signed and dated written informed consent prior to study participation.
8. Normal electrocardiogram (ECG) with QTc <450 msec.
9. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia).
5. Subjects with a family history of sudden cardiac death.
6. A creatinine clearance <70 mL/min as determined by Salazar- Corcoran equations For men : [ 137- age]x [ ( 0.285x weight(kg0) +( 12.1x height(m)2]/ (51xSCr). For women; [146 - age]x( 0.287xweight(kg))+( 9.74xheight(m)2]/(60xSCr)

   Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Salazar, 1988].
7. History of alcohol or substance abuse or dependence within 6 months of the study: History of regular alcohol consumption averaging >7 drinks/wk for women or >14 drinks/wk for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits within 6 months of screening.
8. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
9. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
10. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample.
11. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
12. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. Subjects with unstable medical conditions that, in the opinion of the investigator would compromise their participation in the trial.
13. Subjects with unstable medical conditions that, in the opinion of the investigator would compromise their participation in the trial.
14. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
15. Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
16. AST or ALT >1.5 upper limit of normal (ULN)
17. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
18. G6PD deficient.
19. Abnormal methaemoglobin level. (Normal range 0-3%)
20. History of malaria treatment with Primaquine within 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time AUC 0-∞curve for primaquine and metabolites (mPQ) | 24 hours

SECONDARY OUTCOMES:
Metabolites (mPQ) maximum concentrations (Cmax) of Primaquine | 24 hours
Metabolites (mPQ) elimination rate constants (mPQ-λz) | 24 hours
Elimination half life (mPQ-t1/2) of Primaquine | 24 hours
Number of adverse events (Safety and tolerability) | 48 hours
  adverse events, clinical laboratory and vital signs assessments will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes